CLINICAL TRIAL: NCT04773444
Title: Effects of Eccentric and Concentric Cycling Exercise Regimens on Hemodynamic and Hemorheologic Properties in Sedentary Male
Brief Title: Eccentric Cycling Exercise on Hemodynamic and Hemorheologic Properties
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jong-Shyan Wang, Consultant, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201900415A3C
Record Dates: First submitted 2021-02-25; First posted 2021-02-26 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Eccentric Exercise Training
Keywords: eccentric cycling; erythrocyte; hemodynamic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eccentric cycling training (Experimental): Moderate intensity cycling training in eccentric type
  Interventions: Behavioral: Eccentric cycling training
- Concentric cycling training (Experimental): Moderate intensity cycling training in concentric type (intensity matched the eccentric training)
  Interventions: Behavioral: Concentric cycling training
- Control group (No Intervention): without receiving any exercise training

INTERVENTIONS:
Behavioral: Eccentric cycling training — 1. Performed exercise training 5 days a week for 6 weeks on an eccentric ergometer.
  2. Each training session: 3 min at 30% of maximal workload (Wmax) for warmed up and cold down and 30 min the main training phase.
  3. Intensity: Firstly, set at 45% Wmax, and progressively increased 5% per week
  Arms: Eccentric cycling training
Behavioral: Concentric cycling training — 1. Performed exercise training 5 days a week for 6 weeks on an eccentric ergometer.
  2. Each training session: 3 min at 30% of maximal workload (Wmax) for warmed up and cold down and 30 min the main training phase.
  3. Intensity: Firstly, set at 45% Wmax, and progressively increased 5% per week
  Arms: Concentric cycling training

SUMMARY:
The effects of an eccentric endurance training on central and peripheral hemodynamic adaptations and erythrocyte rheology during maximal exercise remained to be unexplored. The current study examined the contribution of rheological functions and/or hemodynamic adaptation to changes in oxygen consumption (VO2) following the matched-power output eccentric (ECT) or concentric cycling training (CCT).

Method: A total of 39 sedentary males were randomly assigned into either CCT (n=13) or ECT (n=13) for 30 min a day, 5 days a week for 6 weeks at 60% of maximal workload or to a CTL (control group, n = 13). A graded exercise test (GXT) was performed before and after the intervention. Central and microvascular adaptations were evaluated using thoracic impedance and near-infrared spectroscopy (NIRS), respectively. Rheological characteristics was determined by an ektacytometer.

DETAILED DESCRIPTION:
Endurance training is a well known strategy for improving fitness capacity. However, some populations are intolerance to complete the usual exercise training program, such as chronic heart or pulmonary disease or the elderly. Therefore, ECT is a candidate training strategy for those individuals.

Erythrocytes deformability is significantly related to the blood perfusion in microcirculation. The impaired erythrocyte-related rheology further lead to reduced aerobic capacity by our research team. Therefore, the lower energy consumed in ECT may avoid the oxidative stress. To now, less studies have demonstrated whether ECT influences peripheral hemodynamics by erythrocyte rheology and the blood flow from the central effect.

The investigators aimed to investigate the effects of CCT and ECT on oxygen consumption response explained by changes in local blood perfusion, blood cell rheology, or central function to attempt developing its application in rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* in sedentary lifestyle, who were nonsmokers, nonusers of medications/vitamins, and free of any cardiopulmonary/hematological risks

Exclusion Criteria:

* regular exercise habits (i.e., exercise frequency once per week, duration >20 min).

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-11 (Actual); Primary Completion 2022-05-16 (Estimated); Study Completion 2022-05-16 (Estimated)

PRIMARY OUTCOMES:
Central and peripheral hemodynamics | 12 weeks
  Evaluate cardiac and peripheral hemodynamic response to exercise by using noninvasive continuous cardiac output monitoring system and near-infrared spectroscopy (NIRS).

SECONDARY OUTCOMES:
Cardiopulmonary fitness | 12 weeks
  The graded exercise test (GXT) on a bicycle ergometer was performed. The GXT comprised 2 min of unloaded pedaling followed by a continuous increase in the work rate of 30 watt per 3-minute until exhaustion (i.e., progressive exercise to maximal O2 consumption)
Erythrocyte rheological characteristics | 12 weeks
  Isolated erythrocyte first, then detect the cell geometric shape by using the FACSCalibur.
  To assess erythrocyte deformability and aggregation by using laser assisted optical rotational red cell analyzer (LoRRca).

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Shyan Wang, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoppeler H. Moderate Load Eccentric Exercise; A Distinct Novel Training Modality. Front Physiol. 2016 Nov 16;7:483. doi: 10.3389/fphys.2016.00483. eCollection 2016. PMID 27899894
- [Background] Haynes A, Linden MD, Chasland LC, Nosaka K, Maiorana A, Dawson EA, Dembo LH, Naylor LH, Green DJ. Acute impact of conventional and eccentric cycling on platelet and vascular function in patients with chronic heart failure. J Appl Physiol (1985). 2017 Jun 1;122(6):1418-1424. doi: 10.1152/japplphysiol.01057.2016. Epub 2017 Mar 16. PMID 28302709
- [Background] Lindstedt SL, LaStayo PC, Reich TE. When active muscles lengthen: properties and consequences of eccentric contractions. News Physiol Sci. 2001 Dec;16:256-61. doi: 10.1152/physiologyonline.2001.16.6.256. No abstract available. PMID 11719600
- [Result] LaStayo PC, Ewy GA, Pierotti DD, Johns RK, Lindstedt S. The positive effects of negative work: increased muscle strength and decreased fall risk in a frail elderly population. J Gerontol A Biol Sci Med Sci. 2003 May;58(5):M419-24. doi: 10.1093/gerona/58.5.m419. PMID 12730250